CLINICAL TRIAL: NCT03954587
Title: What is the Optimal Cycle Regimen for Frozen- Thawed Embryo Transfer Cycles: Spontaneous Natural Cycles Versus Hormonal Replacement Treatment (HRT) Cycles
Brief Title: What is the Optimal Cycle Regimen for Frozen- Thawed Embryo Transfer Cycles
Status: Terminated | Type: Observational
Why Stopped: Investigator's perogative
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Prof Dr. Human Fatemi, Medical Director, ART Fertility Clinics LLC
Other Study IDs: 1901-ABU-015-CC
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Infertility; Female Infertility; Pregnancy Early
Keywords: Hormone replacement therapy; Frozen thawed embryos; Frozen embryo cycle
MeSH Terms: conditions — Infertility; Infertility, Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Artificial (HRT) Cycles: 1. Commence estradiol valerate (E2) 4mg from day 2 or 3 of period for 3 days
  2. Increase E2 to 6mg on day 4 of E2 treatment, according to clinician discretion based on endometrial thickness.
  3. Transvaginal scan throughout the HRT cycle to not only monitor endometrial development but to also exclude the presence of a dominant follicle on the ovaries.
  4. Serial measurements of serum LH (luteinizing hormone), estradiol and progesterone levels.
  5. Initial progesterone dose of 100mg at 22hrs (vaginal suppository) after ≥ 7 days and ≤ 16 days of estradiol administration when the minimal endometrial thickness achieved is 6mm with a trilaminar appearance.
  6. Subsequently increase progesterone administration to 100mg vaginally three times daily. Continue E2 administration 6mg (3 tablets daily).
  7. Embryo transfer is scheduled on the 5th full day of progesterone administration.
- Spontaneous natural cycles:: 1. Day 2 of menses and throughout patients' natural cycle scans to monitor follicular growth.
  2. Measurements of serum LH, estradiol and progesterone levels to determine ovulation.
  3. The LH surge will be considered to have begun when the concentration rises by 180% above the most recent serum value and continues to rise thereafter (Irani et al. 2017, Fatemi et al., 2010).
  4. Day 1 after the LH rise, a decrease in estradiol concentration is identified. Twenty four hours later progesterone concentrations rise with a level of greater than or equal to 1.5ng/mL confirming ovulation (day 0) (Irani et al., 2017; Speroff et al.). This is considered as day 0 with initiation of vaginal progesterone 100mg at 22hrs that night. The following day (day 1) the patient increases progesterone administration to 100mg vaginally 8 hourly and continues until 7 weeks gestation as per clinic protocol. Embryo transfer is scheduled 5 days (day 5) following confirmation of ovulation (day 0).

SUMMARY:
Investigators will be comparing artificial (HRT) frozen-thawed embryo transfer cycles to correctly conducted spontaneous natural cycles after the transfer of a chromosomally normal embryo.

DETAILED DESCRIPTION:
The most common treatment protocols for frozen embryo transfers include natural cycles with or without human chorionic gonadotrophin (HCG) trigger or endometrial preparation with hormonal treatment (artificial cycles), with or without Gonadotrophin - releasing hormone agonist suppression. Recent studies comparing artificial and natural cycles concluded that the optimal means of endometrial preparation for frozen- thawed cycle remains unclear and both options may be offered to women with regular ovulatory cycles.

Correctly identified spontaneous natural cycles are the preferred option for frozen-thawed embryo transfer in women with regular menstrual cycles.

Investigators will be comparing artificial (HRT) frozen-thawed embryo transfer cycles to correctly conducted spontaneous natural cycles after the transfer of a chromosomally normal embryo.

ELIGIBILITY:
Inclusion criteria include the following:

1. Women aged 18 years to 42 years with regular menses (26-34 days)
2. Having 1 or 2 chromosomally normal cryopreserved blastocysts available for transfer.
3. First frozen-thawed transfer cycle
4. Progesterone level < 1.5 ng/mL day of trigger injection in stimulation cycle from which embryos to be transferred were created.

Exclusion criteria include the following:

1. Polycystic ovarian syndrome
2. Poor ovarian responder in accordance with Bologna criteria
3. Uterine abnormality US / saline infusion sonohysterogram
4. Previous dilatation & curettage (D&C)
5. Hydrosalpinx
6. Asherman syndrome
7. History of endometriosis
8. ICSI due to severe male factor with testicular sperm
9. Any known contraindications or allergy to oral estradiol or progesterone.
10. Discontinuation of HRT medication ( medication error in research HRT cycle )
11. Failure to detect ovulation in the research natural cycle
12. Duration of estradiol exposure ≥ 17 days and endometrium < 6mm
13. Spontaneous ovulation in HRT artificial cycle

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female under infertility treatment
Study Population: Female who underwent a previous ovarian stimulation for In Vitro Fertilisation/Intracytoplasmic Sperm Injection with pre-implantation genetic screening and embryo vitrification, who are planned for their first frozen thaw embryo transfer cycle
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate to 8 weeks gestation | 8 weeks
  viable pregnancy to 8 gestational weeks
Pregnancy rate beta human chorionic gonadotropin (ß-hCG) > 5 IU | 12 days
  Number of patients with a hCG > 5 IU out of the number of patients who underwent an embryo transfer with one or two euploid embryos
Biochemical pregnancy rate | 5 weeks
  Positive ß-hCG, but at 5 gestational weeks no ultrasonographic visible gestational sac seen
Clinical implantation rate | 6 weeks
  Number of gestational sacs observed by ultrasound at 6 weeks of gestation divided by the number of embryos transferred
Clinical pregnancy rate | 5 weeks
  Ultrasonographic visible sac at 5 gestational weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carol Coughlan, PhD, Principal Investigator — IVI Middle East Fertility Clinic LLC
Locations (1):
- IVI Middle East Fertility Clinic, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roque M, Lattes K, Serra S, Sola I, Geber S, Carreras R, Checa MA. Fresh embryo transfer versus frozen embryo transfer in in vitro fertilization cycles: a systematic review and meta-analysis. Fertil Steril. 2013 Jan;99(1):156-162. doi: 10.1016/j.fertnstert.2012.09.003. Epub 2012 Oct 3. PMID 23040524
- [Background] Roque M, Valle M, Guimaraes F, Sampaio M, Geber S. Freeze-all policy: fresh vs. frozen-thawed embryo transfer. Fertil Steril. 2015 May;103(5):1190-3. doi: 10.1016/j.fertnstert.2015.01.045. Epub 2015 Mar 4. PMID 25747130
- [Background] Bourgain C, Devroey P. The endometrium in stimulated cycles for IVF. Hum Reprod Update. 2003 Nov-Dec;9(6):515-22. doi: 10.1093/humupd/dmg045. PMID 14714588
- [Background] Devroey P, Bourgain C, Macklon NS, Fauser BC. Reproductive biology and IVF: ovarian stimulation and endometrial receptivity. Trends Endocrinol Metab. 2004 Mar;15(2):84-90. doi: 10.1016/j.tem.2004.01.009. PMID 15036255
- [Background] Kolibianakis E, Bourgain C, Albano C, Osmanagaoglu K, Smitz J, Van Steirteghem A, Devroey P. Effect of ovarian stimulation with recombinant follicle-stimulating hormone, gonadotropin releasing hormone antagonists, and human chorionic gonadotropin on endometrial maturation on the day of oocyte pick-up. Fertil Steril. 2002 Nov;78(5):1025-9. doi: 10.1016/s0015-0282(02)03323-x. PMID 12413988
- [Background] Nikas G, Develioglu OH, Toner JP, Jones HW Jr. Endometrial pinopodes indicate a shift in the window of receptivity in IVF cycles. Hum Reprod. 1999 Mar;14(3):787-92. doi: 10.1093/humrep/14.3.787. PMID 10221715
- [Background] Simon C, Garcia Velasco JJ, Valbuena D, Peinado JA, Moreno C, Remohi J, Pellicer A. Increasing uterine receptivity by decreasing estradiol levels during the preimplantation period in high responders with the use of a follicle-stimulating hormone step-down regimen. Fertil Steril. 1998 Aug;70(2):234-9. doi: 10.1016/s0015-0282(98)00140-x. PMID 9696213
- [Background] Weinerman R, Mainigi M. Why we should transfer frozen instead of fresh embryos: the translational rationale. Fertil Steril. 2014 Jul;102(1):10-8. doi: 10.1016/j.fertnstert.2014.05.019. Epub 2014 Jun 2. PMID 24890274
- [Background] Liu Y, Lee KF, Ng EH, Yeung WS, Ho PC. Gene expression profiling of human peri-implantation endometria between natural and stimulated cycles. Fertil Steril. 2008 Dec;90(6):2152-64. doi: 10.1016/j.fertnstert.2007.10.020. Epub 2008 Jan 14. PMID 18191855
- [Background] Haouzi D, Assou S, Mahmoud K, Tondeur S, Reme T, Hedon B, De Vos J, Hamamah S. Gene expression profile of human endometrial receptivity: comparison between natural and stimulated cycles for the same patients. Hum Reprod. 2009 Jun;24(6):1436-45. doi: 10.1093/humrep/dep039. Epub 2009 Feb 26. PMID 19246470
- [Background] Ghobara T, Gelbaya TA, Ayeleke RO. Cycle regimens for frozen-thawed embryo transfer. Cochrane Database Syst Rev. 2017 Jul 5;7(7):CD003414. doi: 10.1002/14651858.CD003414.pub3. PMID 28675921
- [Background] Groenewoud ER, Cantineau AE, Kollen BJ, Macklon NS, Cohlen BJ. What is the optimal means of preparing the endometrium in frozen-thawed embryo transfer cycles? A systematic review and meta-analysis. Hum Reprod Update. 2013 Sep-Oct;19(5):458-70. doi: 10.1093/humupd/dmt030. Epub 2013 Jul 2. PMID 23820515
- [Background] Groenewoud ER, Cohlen BJ, Macklon NS. Programming the endometrium for deferred transfer of cryopreserved embryos: hormone replacement versus modified natural cycles. Fertil Steril. 2018 May;109(5):768-774. doi: 10.1016/j.fertnstert.2018.02.135. PMID 29778369
- [Background] Agha-Hosseini M, Hashemi L, Aleyasin A, Ghasemi M, Sarvi F, Shabani Nashtaei M, Khodarahmian M. Natural cycle versus artificial cycle in frozen-thawed embryo transfer: A randomized prospective trial. Turk J Obstet Gynecol. 2018 Mar;15(1):12-17. doi: 10.4274/tjod.47855. Epub 2018 Mar 29. PMID 29662710
- [Background] Fatemi HM, Kyrou D, Bourgain C, Van den Abbeel E, Griesinger G, Devroey P. Cryopreserved-thawed human embryo transfer: spontaneous natural cycle is superior to human chorionic gonadotropin-induced natural cycle. Fertil Steril. 2010 Nov;94(6):2054-8. doi: 10.1016/j.fertnstert.2009.11.036. Epub 2010 Jan 25. PMID 20097333
- [Background] Zimmermann G, Ackermann W, Alexander H. Epithelial human chorionic gonadotropin is expressed and produced in human secretory endometrium during the normal menstrual cycle. Biol Reprod. 2009 May;80(5):1053-65. doi: 10.1095/biolreprod.108.069575. Epub 2009 Jan 21. PMID 19164178
- [Background] Shi Y, Sun Y, Hao C, Zhang H, Wei D, Zhang Y, Zhu Y, Deng X, Qi X, Li H, Ma X, Ren H, Wang Y, Zhang D, Wang B, Liu F, Wu Q, Wang Z, Bai H, Li Y, Zhou Y, Sun M, Liu H, Li J, Zhang L, Chen X, Zhang S, Sun X, Legro RS, Chen ZJ. Transfer of Fresh versus Frozen Embryos in Ovulatory Women. N Engl J Med. 2018 Jan 11;378(2):126-136. doi: 10.1056/NEJMoa1705334. PMID 29320646
- [Background] O'Connor KA, Brindle E, Miller RC, Shofer JB, Ferrell RJ, Klein NA, Soules MR, Holman DJ, Mansfield PK, Wood JW. Ovulation detection methods for urinary hormones: precision, daily and intermittent sampling and a combined hierarchical method. Hum Reprod. 2006 Jun;21(6):1442-52. doi: 10.1093/humrep/dei497. Epub 2006 Jan 26. PMID 16439502
- [Background] Irani M, Robles A, Gunnala V, Reichman D, Rosenwaks Z. Optimal parameters for determining the LH surge in natural cycle frozen-thawed embryo transfers. J Ovarian Res. 2017 Oct 16;10(1):70. doi: 10.1186/s13048-017-0367-7. PMID 29037231